CLINICAL TRIAL: NCT00535080
Title: Compassionate Use of Metvix® (Methyl Aminolevulinate) PDT in Subjects With Field Actinic Keratoses, Large/Multiple Superficial BCCs, or Bowen's Disease
Brief Title: Compassionate Use of Metvix® (Methyl Aminolevulinate) Photodynamic Therapy (PDT) in Subjects With Field Actinic Keratoses, Large/Multiple Superficial Basal Cell Carcinomas (BCCs), or Bowen's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Galderma R&D (Industry)
Responsible Party: Director, Regulatory, Medical & Technical Affairs, Galderma Canada
Other Study IDs: CAN.15.SPR.001
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2009-10

CONDITIONS: Field Actinic Keratoses; Basal Cell Carcinoma; Bowen's Disease
Keywords: actinic; keratoses; superficial; basal; carcinomas; Bowen's; large or multiple superficial Basal Carcinomas
MeSH Terms: conditions — Carcinoma, Basal Cell; Bowen's Disease; Keratosis; Carcinoma | interventions — methyl 5-aminolevulinate

INTERVENTIONS:
Drug: Metvix (methyl aminolevulinate) — Metvix (methyl aminolevulinate) (MAL), Photodynamic Therapy (PDT), cream, 160 mg/g. MAL cream will be applied for 3 hours then will be removed. The target area will then be exposed to red light (using a large-field LED light source: Aktilite 128) for 7 to 10 minutes at a dosage of 37 J/cm².

SUMMARY:
The aim of this study is to provide this investigational drug to patients who cannot be optimally treated with conventional therapies and to collect efficacy and safety data on the use of Metvix PDT in subjects with field actinic keratoses, large/multiple superficial basal cell carcinomas (BCCs) or Bowen's disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject older than 18 years.
* Subject presenting with:

  * Either field actinic keratoses (AKs) (mild to moderate, multiple and clustered AKs on a severely sun-damaged skin); or
  * Biopsy-confirmed large, or multiple (several in the same anatomical area) primary superficial BCC lesions that are macroscopically and histologically consistent with superficial basal cell carcinoma (sBCC) and have no histological evidence of aggressive growth patterns; or
  * Histologically confirmed diagnosis of Bowen's disease from a biopsy taken within 3 months
* Any subject presenting with the aforementioned lesions must not be able to be treated optimally by conventional therapies.
* Female subject of childbearing potential, using an effective birth control method (see Case Report Form) and having a negative pregnancy test at the beginning of the study, or female subject of non childbearing potential
* Subject must be willing and capable of cooperating to the extent and degree required by the protocol.
* Subject has to read Patient Information Sheet and read and sign the Informed Consent form prior to any study related procedure.

Exclusion Criteria:

* A recurrent superficial BCC lesion that has previously been treated.
* Subject whose lesions on the selected treatment zone (including a 5 cm margin around the treatment area) have been treated with any of the following topical treatments within the specified washout period:

  * 5-FU - 3 months
  * Cryotherapy - 3 months
  * Imiquimod - 3 months
  * PDT - 3 months
  * Diclofenac sodium - 3 months
  * Surgery, radiotherapy, curettage, electrodesiccation, retinoids, dermabrasion, laser resurfacing, salicylic acid - 3 months
* A primary superficial BCC located close to or involving a scar of SCC
* Subject with known porphyria.
* Subject with target lesions on the genitals.
* Subject with known xeroderma pigmentosum.
* Pigmented lesion(s) on the treated area.
* Morpheaform lesion(s) on the treated area.
* Infiltrating lesion(s) on the treated area.
* Female subject who is pregnant, nursing or planning a pregnancy during the study.
* Subject with known hypersensitivity to methyl 5-aminolevulinate, a similar compound or excipients of the cream.
* Subject who has participated in another investigational drug or device research study within 30 days of enrolment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Related Info — http://www.galderma.com/